CLINICAL TRIAL: NCT02505386
Title: Pharmacokinetics of Ertapenem Following Subcutaneous or Intravenous Infusion in Patients Aged Over 75 (PHACINERTA)
Brief Title: Pharmacokinetics of Ertapenem in Patients Aged Over 75
Acronym: PHACINERTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHUBX 2013/12
Record Dates: First submitted 2014-08-04; First posted 2015-07-22 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Infections
Keywords: Ertapenem; Subcutaneously; Aged; Elderly; Pharmacokinetics
MeSH Terms: conditions — Infections | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ertapenem IV (Active Comparator): IV administration of ertapenem
  Interventions: Drug: Ertapenem
- Ertapenem SC (Experimental): SC administration of ertapenem
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem

SUMMARY:
In geriatric departments, physicians are faced with two difficulties, first the increasing number of infections caused by multiresistant bacteria, especially extended spectrum β-lactamase (ESBL) producing enterobacteria strains and second, the poor venous access frequently encountered in elderly population. Giving antibiotics subcutaneously would be an interesting alternative, all the more as intramuscular injection is contraindicated in case the of anticoagulant therapy. Unfortunately, few data are available about subcutaneous (SC) administration. Ertapenem is a recent long-acting parenteral carbapenem indicated especially in the treatment of ESBL infection. Its subcutaneously administration has been tested in several studies in Intensive Care Units (ICU) and internal medicine wards with promising results regarding clinical and pharmacokinetics data.

An alternative to the IV Ertapenem administration is needed because of poor venous access and behavioural abnormalities commonly present in infected elderly population. Ertapenem is currently SC administrated in geriatric departments if no other option is available. Moreover elderly patients often present several comorbdities, polymedication, renal insufficiency, cachexia which may disturb antibiotics pharmacokinetics.

The aim of the study is to obtain pharmacokinetic data of SC and IV Ertapenem administration in elderly population, obtain PK/PD parameters adapted to time-dependent antibiotics (T%>MIC) and descriptive data of occurrence of adverse effects and evolution of signs of infection.

DETAILED DESCRIPTION:
ESBL infection incidence increases especially in elderly population (Observatoire National de l'Epidémiologie de la Résistance Bactérienne aux Antibiotiques (ONERBA) www.onerba.org). SC antibiotic route is sometimes the only option available for infected elderly patients (delirium, dementia or no venous access) and presents advantages like greater patient comfort, less nursing time and decrease hospital duration. Ertapenem has a relatively long half life (4 hours) compared to imipenem (1 hour) and a less broad spectrum. Two studies compared the ertapenem pharmacokinetics regarding IV or SC administration. The first concerned 6 patients admitted in ICU and the second 16 patients in internal medicine department. They found IV and SC administrations were equivalent considering that ertapenem antimicrobial activity was time dependent. In fact, a reduction of peak concentration and of time to peak concentration was observed in both studies, but the Area Under the Curve were similar especially the time spent over the Minimal Inhibitory Concentration. Both studies did not observe any severe adverse effects. Because of these promising results and despite not being approved yet, SC Ertapenem, is commonly used in geriatric department. This administration route is chosen when no other option is available, for instance in cases of behavioural disturbance and lack of venous access.

The objective of the investigators study is to confirm the pharmacokinetics data in elderly population known to present frequently renal insufficiency and denutrition and to document the occurrence of adverse effects and clinical evolution.

Patients over 75 receiving ertapenem for 48 hours (IV or SC) will be included. Ertapenem concentrations (H0, H+0.5h and H+2.5h) will be determined at steady state and described based on administration route. Systemic and local adverse effects will be collected during the treatment and infection evolution will be described.

Patients will be monitored during ertapenem treatment and for 45 days after the beginning of the treatment. Biological data will be obtained initially at inclusion (D3 after ertapenem beginning) and for 14 days (+/-10) after the beginning of the treatment (corresponding to end of treatment). Signs of infection evolution will be also monitored for 45 days (+/-10).

ELIGIBILITY:
Inclusion Criteria:

* Age> or equal to 75 years
* Treatment with ertapenem (1g daily) for at least 48 hours IV or SC (or one then the other)
* Subject affiliated or beneficiary of a social security system,
* Free Consent, informed and signed by the participant or by the designation of a proxy if delirium and the investigator.

Exclusion Criteria:

* Age < 75 years
* Criteria for legislation: those under protection of the justice, subject participating in other research, including a period of exclusion still going to pre-inclusion

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve established from the minimal concentration | 48 hours after ertapenem beginning
  To determine and compare Area under the curve established from the minimal concentration, Maximal concentration n°1 (at the end of the infusion) and Maximal concentration n°2 (2 hours after the end of the infusion) between intravenous and subcutaneous (SC) routes

SECONDARY OUTCOMES:
Time spent over the minimal inhibitory concentration | 48 hours after ertapenem beginning
  To assess the time spent over the minimal inhibitory concentration
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | From the ertapenem beginning until 15 days after the end of the treatment
  To assess and graduate the number of AE
Proportion of recovery | At the end of the treatment
  To assess the efficacy of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claire ROUBAUD BAUDRON, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Roubaud Baudron C, Legeron R, Ollivier J, Bonnet F, Greib C, Guerville F, Cazanave C, Kobeh D, Cressot V, Moneger N, Videau MN, Thiel E, Foucaud C, Lafargue A, de Thezy A, Durrieu J, Bourdel Marchasson I, Pinganaud G, Breilh D. Is the subcutaneous route an alternative for administering ertapenem to older patients? PHACINERTA study. J Antimicrob Chemother. 2019 Dec 1;74(12):3546-3554. doi: 10.1093/jac/dkz385. PMID 31730164